CLINICAL TRIAL: NCT07295808
Title: Identification and Characterisation of IgA With Nephritogenic Potential in IgA Deposition Nephropathies
Brief Title: Identification and Characterisation of IgA With Nephritogenic Potential in IgA Deposition Nephropathies (Rep-IgAN)
Acronym: Rep-IgAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI24_0003 - Rep-IgAN
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Kidney Disease
Keywords: Kidney disease; Immunoglobulin A; Berger's disease
MeSH Terms: conditions — Kidney Diseases; Glomerulonephritis, IGA | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample taken in a Tempus tube during a blood test performed at the same time as the kidney bio (Other): Blood sample taken in a Tempus tube during a blood test performed at the same time as the kidney biopsy.
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample taken in a Tempus tube during a blood test performed at the same time as the kidney biopsy.

SUMMARY:
IgA nephropathy (IgA Nephropathy), or Berger's disease, is the most common form of primary glomerulonephritis. It is a major cause of end-stage renal failure, often leading to dialysis or kidney transplantation. Recurrence is common after transplantation, compromising graft survival. Rheumatoid purpura (or IgA vasculitis) shares a common pathophysiology with IgA N, characterised by mesangial deposits containing IgA-rich immune complexes, but differs in its systemic involvement (skin, joints and digestive system).

In terms of pathophysiology, the histological signature of these conditions is based on the accumulation of abnormal IgA within the glomerulus. The mechanisms responsible for the nephrotoxicity of these IgA remain partially unclear. In patients with NIgA, several qualitative abnormalities of IgA have been well described, including a glycosylation defect that promotes IgA polymerisation and the emergence of anti-IgA autoantibodies. These immune complexes, found in glomerular deposits, induce a local inflammatory reaction. Experimental work conducted on mouse models developed at the CRIBL laboratory has shown that these abnormalities may be linked to a dysregulation of the immune response, leading to the production of IgA with physicochemical properties that promote their deposition in the kidney.

However, the location of nephritogenic IgA-secreting B cells remains poorly understood. Recent data suggest that this production could occur directly within the renal parenchyma, where activated B lymphocytes would locally produce pathogenic IgA. Following on from these observations, our study aims to characterise the immunoglobulin (Ig) repertoires in patients with IgA nephropathy, particularly those from renal lymphoid infiltrates, and to compare them with the repertoires of circulating B cells.

We hypothesise that certain sequence motifs within the variable domains of IgA, particularly the CDR3 regions, could constitute specific biomarkers of NIgA. Their detection in peripheral blood could enable non-invasive or predictive diagnosis, complementing the renal biopsy that is currently essential.

ELIGIBILITY:
Inclusion Criteria:

* Patients of interest: all patients with IgA nephropathy or rheumatoid purpura aged 18 years or older whose treatment requires a renal biopsy
* Control patients: all patients with a renal disease other than IgA nephropathy or rheumatoid purpura whose treatment requires a renal biopsy

Exclusion Criteria:

* Patient opposition
* Persons under legal guardianship
* Persons whose psychological health prevents the collection of non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2029-06-25 (Estimated); Study Completion 2029-07-25 (Estimated)

PRIMARY OUTCOMES:
Variable domains of IgA | 6 months
  Describe the repertoire of variable domains of IgA with nephritogenic potential in patients with IgA nephropathies

SECONDARY OUTCOMES:
Direct in situ lymphoid infiltrate mapping within the kidney | 6 months
  Search circulating repertoires, based on a blood sample taken at the time of diagnosis and at the same time as the renal biopsy, for the presence of nephritogenic IgA previously identified using the renal Ig repertoire.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No